CLINICAL TRIAL: NCT00729599
Title: Single Site Study, Phase III, for Safety Dermatological Evaluation: Basic Acceptability With Odontological Follow up - Cepacol Teen.
Brief Title: Safety Dermatological Evaluation: Acceptability With Odontological Follow up - Cepacol Teen.
Acronym: Cepacol Teen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPYRY_L_04020
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-03

CONDITIONS: Hygiene
MeSH Terms: interventions — Cetylpyridinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cetylpyridinium chloride during 21 consecutive days.
  Interventions: Drug: Cetylpyridinium chloride

INTERVENTIONS:
Drug: Cetylpyridinium chloride — Cetylpyridinium chloride during 21 consecutive days.

SUMMARY:
To prove the safety, in normal conditions, of the Cepacol Teen, a formulation to odontological usage.

ELIGIBILITY:
Inclusion Criteria:

* Integral buccal mucous (without oral pathologies);
* Normal odontological exams;

Exclusion Criteria:

* Lactation or gestational risk or gestation;
* Use of Antiinflammatory or immunosuppression drugs 15 days before the study;
* Being in odontological treatment;
* Pathological or mucous disease which can interfere or active gynaecological disease which may interfere wtih study results;
* Personal history of allergic disease in the area to be treated;
* Allergic or atopic history;

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Patients will be evaluated according to the adverse reactions and the intensity of them. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, MD, Study Director — Sanofi-aventis administrative office Brazil
Locations (1):
- Sanofi-aventis, São Paulo, São Paulo, Brazil